CLINICAL TRIAL: NCT00395317
Title: Randomised, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study to Investigate the MRI Efficacy and the Safety of Six Months Administration of SB-683699 in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Study Of SB-683699 Compared To Placebo In Subjects With Relapsing-Remitting Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4M105038
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Sclerosis
Keywords: magnetic resonance imaging; multiple sclerosis; SB-683699
MeSH Terms: conditions — Multiple Sclerosis | interventions — Firategrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Placebo Comparator): placebo (4 tablets)
  Interventions: Other: Placebo
- Arm 2 (Experimental): SB-683699 150 mg bid (1 x 150mg + 3 placebo tablets)
  Interventions: Other: Placebo; Drug: Firategrast 150 mg
- Arm 3 (Experimental): SB-683699 600 mg bid (2 x 300mg + 2 placebo tablets)
  Interventions: Other: Placebo; Drug: Firategrast 300 mg
- Arm 4 (Experimental): SB-683699 900 mg bid (3 x 300 mg + 1 placebo tablet)
  Interventions: Other: Placebo; Drug: Firategrast 300 mg
- Arm 5 (Experimental): SB-683699 1200 mg bid, male subjects only (4 x 300 mg tablets)
  Interventions: Drug: Firategrast 300 mg

INTERVENTIONS:
Other: Placebo — placebo tablet
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: Firategrast 150 mg — 150 mg tablet
  Other Names: SB-683699
  Arms: Arm 2
Drug: Firategrast 300 mg — 300 mg tablet
  Other Names: SB-683699
  Arms: Arm 3; Arm 4; Arm 5

SUMMARY:
SB-683699 is an oral medication that is thought to reduce the number of active white blood cells entering the brain; these white blood cells are part of the disease process for MS. This study will look at whether different doses of SB-683699 are effective and safe in patients with relapsing remitting MS.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Males or females, aged 18 to 65, inclusive
* A diagnosis of relapsing-remitting MS [Polman, 2005; McDonald, 2001] with dissemination in time and space
* EDSS of between 0 and 6.0 inclusive at the Screening visit
* Occurrence of at least two relapses in previous 24 months with at least one relapse or documented evidence of gadolinium-enhancement on MRI (prior to screening) in the previous 12 months. Subject must not have had a relapse within 4 weeks prior to Screening. In addition, subjects experiencing a relapse between Screen and Visit 3 will not be eligible to be randomized.
* A minimum of five T2 lesions on brain MRI at Visit 2 as determined by the central MRI analysis reader
* A female subject is eligible to enter the study if she is:

  * Of non-childbearing potential, i.e. women who:
  * have documented evidence of tubal ligation, bilateral oophorectomy or hysterectomy; or
  * are post-menopausal, defined as at least one year without menses in the absence of hormone replacement therapy. In questionable cases, menopausal status will be confirmed by oestradiol and FSH levels consistent with menopause according to local laboratory ranges. Oestrogen-containing hormone replacement therapies are not allowed during the study.
  * Of childbearing potential, has a negative urine pregnancy test at Screening, and agrees to the consistent and correct use of one of the methods of contraception listed below. Subjects will use this contraceptive method for at least one month prior to Screening and should continue to use the same contraceptive method throughout the study until at least 3 days after the last dose of investigational product.
  * Progesterone-only oral contraceptives or implants (inserted at least one month prior to Screening, but not beyond the third successive year following insertion). Oestrogen-containing contraceptives are not allowed during the study.
  * Intra-uterine device (IUD) inserted by a qualified clinician. The IUD must have published data showing that the highest expected failure rate is less than 1% per year.
  * Spermicide in conjunction with either a diaphragm, cervical cap or condom. Male partner sterilization (vasectomy) prior to female subject's entry into the study and is the sole partner for that female subject
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subjects receiving corticosteroids within 4 weeks of Screening for treatment of MS. If non-systemic steroids are being used for other chronic inflammatory conditions, subjects may be included at the discretion of the investigator after discussion with the GSK medical monitor
* Use of an b-interferon product, glatiramer acetate or azathioprine within 3 months of Screening, or use of Mitoxantrone within 12 months of Screening. Subjects who have received other therapies affecting the immune system (such as intravenous immunoglobulin (IVIg), cyclophosphamide, plasmapheresis, or any other immunosuppressive or immunomodulatory treatment) in the past may be included on a case by case basis after discussion with the GSK medical monitor. None of these treatments will be allowed during this study
* Previous exposure to alemtuzumab, natalizumab or firategrast administration, bone marrow transplantation or whole body irradiation
* Subjects with a cardiac pacemaker or any other type of metal implant or with any other contraindication for MRI (including known allergy to gadolinium)
* Use of 4-aminopyridine, rosiglitazone, pioglitazone or any drug that is an inhibitor of or a substrate (with a low therapeutic index) for OATP at Screening.
* Subjects with clinically significant renal laboratory values: subjects with a calculated creatinine clearance <60ml/min (by Cockcroft and Gault) at Screening
* Subjects with local urinalysis findings of 1) proteinuria, defined as ≥1+ protein, on urine dipstick or 2) renal tubular cell casts or 3) ≥5 red blood cells / high power field will be excluded from the study if the result is still present on a repeat urinalysis during the screening period.
* Presence of clinically significant hepatic laboratory values: ALT, AST, GGT > 2.0- times the upper limit of normal (ULN); total bilirubin > 1.5 times the ULN at Screening
* CD4 count <500, CD4:CD8 <1.0 (if result still present on a repeat test during the screening period), JC viremia detected in plasma or white cells, idiopathic CD4/CD8 lymphopenia or secondary lymphopenia at Screening
* Any findings on the MRI of the brain at Visit 2 other than MS, except for benign findings that (in the opinion of the central MRI reading site and local site investigator) require no further evaluation or treatment and do not impact patient's neurological health (e.g., small arachnoid cysts, venous angiomas)
* Current or history of cancer, excluding localized non-melanoma skin cancer
* Uncontrolled or any active bacterial, viral, or fungal infection at Screening. Any previous serious infections should be discussed with the GSK medical monitor (e.g. opportunistic or atypical infections)
* History of tuberculosis (TB) or positive chest X-ray for TB at Screening (prior chest X-ray is acceptable if performed within previous 6 months)
* Known congenital or acquired immunodeficiency
* Any abnormality on 12-lead ECG at Screening which is clinically significant in the opinion of the investigator
* Subjects with positive hepatitis B surface antigen, hepatitis C antibody, or HIV tests at Screening
* Women who are lactating, pregnant (positive pregnancy test at Screening), or planning to become pregnant during the course of the study
* Recent history or suspicion of current drug abuse (including analgesic abuse) or alcohol abuse within the last 6 months prior to Screening
* Use of an investigational drug for condition other than MS within 30 days or five half-lives (whichever is longer) preceding Screening. Prior use of an investigational drug for MS should be discussed with the GSK medical monitor
* Any concurrent illness, disability or clinically significant abnormality (including laboratory tests) that may affect the interpretation of clinical efficacy or safety data or prevent the subject from safely completing the assessments required by the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Cumulative number of new gadolinium-enhancing lesions on monthly MRI scans during the Treatment Phase | Baseline and 24 weeks

SECONDARY OUTCOMES:
Cumulative volume of new gadolinium-enhancing lesions on monthly MRI scans | Baseline and 24 weeks
Cumulative number of persistent gadolinium-enhancing lesions on monthly MRI scans | Baseline and 24 weeks
Cumulative number of total enhancing lesions on monthly MRI scans: the sum of new and persistent gadolinium-enhancing lesions | Baseline and 24 weeks
Cumulative number of new T1 hypointense lesions on MRI scans | Baseline and 24 weeks
Cumulative number of new/newly enlarging T2 lesions on MRI scans | Baseline and 24 weeks
Relapses Occurring during the On-Treatment Phase | Baseline and 24 weeks
Change from Baseline in Expanded Disability Status Scale (EDSS) scores | Baseline and 24 weeks
Change from Baseline in Multiple Sclerosis Functional Composite (MSFC)scores | Baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- Australia (4):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Austria (2):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
- Canada (4):
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
- GSK Investigational Site, Turku, Finland
- France (7):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Strasbourg
- Germany (14):
  - GSK Investigational Site, Neuburg an der Donau, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Herborn, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Honnef, North Rhine-Westphalia
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (5):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Gallarate, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Siena, Tuscany
- Netherlands (6):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Venray
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Wellington
- Norway (5):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Sandnes
  - GSK Investigational Site, Skien
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (6):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- United Kingdom (5):
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Hartshill, Stoke-on-Trent
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Derived] Miller DH, Weber T, Grove R, Wardell C, Horrigan J, Graff O, Atkinson G, Dua P, Yousry T, Macmanus D, Montalban X. Firategrast for relapsing remitting multiple sclerosis: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2012 Feb;11(2):131-9. doi: 10.1016/S1474-4422(11)70299-X. Epub 2012 Jan 5. PMID 22226929